CLINICAL TRIAL: NCT02723279
Title: A Comparison Study on Efficacies of Electrical Pudendal Nerve Stimulation and Tolterodine Tartrate for Urgency-Frequency Syndrome in Women
Brief Title: Comparison of Electrical Pudendal Nerve Stimulation and Tolterodine Tartrate for Urgency-Frequency Syndrome in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201512ZYSUFS
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Urgency-frequency Syndrome
Keywords: Urgency-frequency Syndrome; Electrical Pudendal Nerve Stimulation; Tolterodine Tartrate
MeSH Terms: interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPNS group (Experimental)
  Interventions: Behavioral: EPNS
- TT group (Active Comparator)
  Interventions: Drug: TT

INTERVENTIONS:
Behavioral: EPNS — Electrical pudendal nerve stimulation Four sacral points are selected. The two upper points are located about 1 cm bilateral to the sacrococcygeal joint. On the upper points, a needle of 0.40 Х 100 mm is inserted perpendicularly to a depth of 80 to 90 mm to produce a sensation referred to the urethra or the anus. The locations of the two lower points are about 1 cm bilateral to the tip of the coccyx. On the lower points, a needle of 0.40 Х 100 or 125 mm is inserted obliquely towards the ischiorectal fossa to a depth of 90 to 110 mm to produce a sensation referred to the urethra. After the sensation referred to the above regions is produced, each of two pairs of electrodes from a G6805-2 Multi-Purpose Health Device is connected with the two ipsilaterally inserted needles.
  Other Names: electrical pudendal nerve stimulation
  Arms: EPNS group
Drug: TT — Tolterodine tartrate (GSK， UK) 4mg per day is taken orally for six weeks
  Other Names: Tolterodine tartrate
  Arms: TT group

SUMMARY:
The purpose of this study is to compare the efficacy of electrical pudendal nerve stimulation (EPNS) and Tolterodine Tartrate in patients with urgency-frequency syndrome.

DETAILED DESCRIPTION:
Tolterodine Tartrate is one of the first-line medications in treatment of Urgency-frequency syndrome (UFS) patients. It is reported to reduce frequency urgency and nocturia and urinary leakage in patients with UFS. However dry mouth and constipation are the most frequently reported adverse events. In other reports blurred vision and increased heart rate are also reported. The side effects limit its application.

Electrical neuromodulation has proved to be valuable in patients with UFS with little adverse effect. The investigators have previously reported electrical pudendal nerve stimulation (EPNS) alone has long term effect in treatment of UFS in women patients. EPNS is developed by combining the advantages of pudendal nerve stimulation (PNS) and percutaneous tibial nerve stimulation (PTNS), and incorporating the technique of deep insertion of long acupuncture needles. Because pudendal nerve (PN) afferents are particularly important for the inhibitory effect on the voiding reflex and SNS only excites part of PN afferents, direct PN stimulation may be more effective. PNS can be used to treat UFS refractory to SNS, but this therapy also has the disadvantages similar to those of SNS. PTNS is minimally invasive, demonstrates efficacy, and is easily applicable and well tolerated, but the results of chronic PTNS treatment are unknown in initially successful patients and PTNS effects diminish over time.

In EPNS, long acupuncture needles of 0.40 Х 100 or 125 mm were deeply inserted into four sacral points and electrified to stimulate the pudendal nerves. CT transverse plane at the coccygeal apex has showed that the position of the lower needle tip is similar to where (adjacent to PN at Alcock's canal) the Bion device is implanted for chronic PN stimulation. Besides the radiographic evidence, simultaneous records of perineal ultrasonographic PFM contraction, vaginal pressure and pelvic floor surface electromyogram in the investigators previous study have proved that EPNS can exactly excite PN. The investigators previous study has also proved that EPNS has a good post-treatment effect on UFS in women. The purpose of the present study is to show the long-term efficacy of EPNS for UFS in women.

ELIGIBILITY:
Inclusion Criteria:

* Urgency with a documented daytime frequency of more than eight voids and/or nocturia of more than one void.

Exclusion Criteria:

* Age <18 years,or >80 years;
* Urinary tract infections based on results of urinalysis or urine culture;
* Painful bladder syndrome manifested by suprapubic pain related to bladder filling accompanied by frequency and other diseases (including interstitial cystitis, neurogenic bladder, bladder tumor, and vesical calculus)
* Causative of urgency and frequency confirmed by physical examination, B-scan ultrasonography.

urodynamic study, cystoscopy, and radiography

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Lower urinary tract syndrome score | 6 weeks
  International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) is used
Quality of life score | 6 weeks
  International Consultation on Incontinence Questionnaire-Quality of life (ICIQ-qol) is used

CONTACTS AND LOCATIONS:
Overall Officials: Siyou Wang, Principal Investigator — Shanghai University of Traditional Chinese Medicine affliated Yueyang Hospital
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided